CLINICAL TRIAL: NCT06257277
Title: Active Surveillance of the Safety of Gadolinium-based Contrast Agent(s) in India
Brief Title: An Observational Study to Collect Information on the Safety of Gadolinium-Based Contrast Agents in Patients in India
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22584
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Contrast Enhancement in Magnetic Resonance Imaging
Keywords: MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients require GBCA-enhanced MRI: Patients who are scheduled to undergo magnetic resonance imaging (MRI) with gadolinium-based contrast agent (GBCA) enhancement as per routine clinical practice.
  Interventions: Drug: GBCAs

INTERVENTIONS:
Drug: GBCAs — GBCAs are given per routine clinical practice.

SUMMARY:
This is an observational study in which data from patients undergoing enhanced MRI using gadolinium based agents (GBCAs) are collected and studied.

An MRI is a test that uses strong magnets and radio waves to make detailed pictures of the inside of the body. The contrast agents commonly used in MRI are gadolinium based contrast agents (GBCAs). GBCAs contain a "rare earth" element called gadolinium (Gd), which helps to increase the signal intensity and contrast in MRI.

GBCAs have been used worldwide for MRI scans. GBCAs are generally considered safe. In some cases, there have been reports of mild to moderate side effects. There have also been reports indicating that small traces of Gd might stay in the body for an extended period after scans. However, there is no clear evidence that this causes any serious or long term problems in patients with normal kidney function.

There are different brands of GBCAs such as Gadovist and Magnevist. Knowledge about the safety of Gadovist and Magnevist in the Indian population is limited.

This study aims to enhance the currently available information on GBCAs and gather more information on the safety of Gadovist and Magnevist in the Indian population during GBCA enhanced MRI procedures in routine practice.

To do this, researchers will collect the following information:

* any possible medical problems occurring immediately after receiving GBCAs (Gadovist and Magnevist), and after 4 and 12 weeks of receiving GBCAs
* frequency of reporting medical problems after the use of GBCAs (Gadovist and Magnevist)

Patients will be asked to take part in the study only after confirming that they need a GBCA enhanced MRI, and the GBCA brand is already identified.

Data will be collected from February 2024 to September 2024. Healthcare professionals will collect safety data from selected sites which frequently conduct GBCA enhanced MRIs for patients who have not received GBCAs before.

Every patient scheduled for an MRI with contrast agents will be followed up at approximately 4 and 12 weeks after the GBCA enhanced MRI.

In this study, only safety data from routine practice are collected.

ELIGIBILITY:
Inclusion Criteria:

* GBCA-naïve male/female patients of at least 18 years of age.
* willing to participate in the active surveillance and agree to be contacted by phone after 6 (±2) weeks after the MR scan for brief interviews.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that require GBCA-enhanced MRI and are willing to participate in the active surveillance and agree to be contacted by phone after 6 (±2) weeks after the MR scan for brief interviews.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Number of adverse events reported after use of branded gadolinium-based contrast agent (GBCA). | Immediately post dose and at 6 (±2) weeks post dose
Number for participants with adverse events after use of a branded GBCA | From injection of GBCAs up to 6 (±2) weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, India

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.